CLINICAL TRIAL: NCT01282190
Title: Effectiveness of Motivational Interview in Patients With Dyslipidemia Treated in Primary Care Consultations (Dislip-EM Study)
Brief Title: Effectiveness of Motivational Interview in Patients With Dyslipidemia
Acronym: Dislip-EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Spanish Society of Family and Community Medicine (Other)
Responsible Party: Principal Investigator, Luis A Perula, Dr, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-0100/2008
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Patients With Dyslipidemia
Keywords: dyslipidemia, motivational interview, prevention
MeSH Terms: conditions — Dyslipidemias | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motivational interview (Experimental)
  Interventions: Behavioral: Motivational interview

INTERVENTIONS:
Behavioral: Motivational interview — Motivational interview

SUMMARY:
Evaluate the effectiveness of motivational interviewing to improve lipid control and cardiovascular risk in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with dyslipidemia
* To sign informed consent.

Exclusion Criteria:

* Secondary hypercholesterolemia.
* Familial hypercholesterolemia.
* Deficiency syndromes family high density lipoprotein.
* Subjects with a history of cardiac or cerebrovascular events.
* Other chronic health problems such as diabetes or severe COPD.
* Subjects with current diagnosis of cancer.
* Patients with hepatic or renal disorders .
* Subjects heavy drinkers.
* Patients with long standing sick leave (more than 6 months).
* Pregnant or breastfeeding.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
lipid levels | 12 months

SECONDARY OUTCOMES:
cardiovascular risk | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Family Medicine Teaching Unit and Community, Córdoba, Córdoba, Spain

REFERENCES:
- [Derived] Boveda-Fontan J, Barragan-Brun N, Campinez-Navarro M, Perula-de Torres LA, Bosch-Fontcuberta JM, Martin-Alvarez R, Arbonies-Ortiz JC, Novo-Rodriguez JM, Criado-Larumbe M, Fernandez-Garcia JA, Martin-Rioboo E; Collaborative Group Estudio Dislip-EM. Effectiveness of motivational interviewing in patients with dyslipidemia: a randomized cluster trial. BMC Fam Pract. 2015 Oct 24;16:151. doi: 10.1186/s12875-015-0370-2. PMID 26498221
- [Derived] Perula LA, Campinez M, Bosch JM, Barragan Brun N, Arbonies JC, Boveda Fontan J, Martin Alvarez R, Prados JA, Martin-Rioboo E, Massons J, Criado M, Fernandez JA, Parras JM, Ruiz-Moral R, Novo JM; collaborative Group Dislip-EM. Is the Scale for Measuring Motivational Interviewing Skills a valid and reliable instrument for measuring the primary care professionals motivational skills?: EVEM study protocol. BMC Fam Pract. 2012 Nov 22;13:112. doi: 10.1186/1471-2296-13-112. PMID 23173902
- [Derived] Perula LA, Bosch JM, Boveda J, Campinez M, Barragan N, Arbonies JC, Prados JA, Martin E, Martin R, Massons J, Criado M, Ruiz R, Fernandez JA, Buitrago F, Olaya I, Perez M, Ruiz J. Effectiveness of Motivational Interviewing in improving lipid level in patients with dyslipidemia assisted by general practitioners: Dislip-EM study protocol. BMC Fam Pract. 2011 Nov 5;12:125. doi: 10.1186/1471-2296-12-125. PMID 22054017
- See also: protocol study — http://www.biomedcentral.com/1471-2296/12/125/abstract